CLINICAL TRIAL: NCT01599221
Title: Observational Retrospective and Prospective Study on the Treatment of Lateral Proximal Femoral Fractures With Medical Device EBA2
Brief Title: Observational Retrospective and Prospective Study on the Treatment of Femoral Fractures With EBA2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Citieffe S.r.l (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: EBA2
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-05

CONDITIONS: Femoral Fractures
Keywords: Femoral fractures; Nail; Implant; Elderly; Orthopaedics
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with EBA2: Subjects who have undergone surgery with EBA2 medical device for lateral proximal femoral fractures
  Interventions: Device: EBA2

INTERVENTIONS:
Device: EBA2 — Surgical implantation of EBA2 medical device in subjects with lateral proximal femoral fractures treated
  Other Names: Endovis B.A.

SUMMARY:
This is an observational, retrospective and prospective study where subjects who have undergone surgery with EBA2 medical device for lateral proximal femoral fractures will be followed for data collection since the day before their surgery (retrospectively) until day 180 after surgery (retrospectively and prospectively).

This study is aimed at collecting data from patients who have already been treated with EBA2 nail. Data collection will cover the details of the fracture and surgery (from which the retrospective nature of the study), as well as details of follow up visits after surgery that patients routinely carry out up to 6 months (from which the prospective nature of the study).

The study will be conducted in three clinical sites in Italy.

DETAILED DESCRIPTION:
EBA2, the technological evolution of Endovis BA, is now available. The device was developed in conformity with Regulations 93/42/CE and 2007/47/CE, it has the CE trademark and it is registered in the Italian National Registry of Medical Devices. EBA2 has the unique features described below:

* it is undersized compared to other nails in commerce, both proximal and distal, to further facilitate the insertion into the bone. The undersizing is aimed to reduce the stiffness of the stem. In particular, the biological nail-bone interaction will be improved as a consequence of lower shear stresses on the frontal plane;
* it is made entirely of titanium. The choice of such a material is aimed to create a flexible means of synthesis that minimizes the differences with the healthy bone mechanical properties and reduces complications in the process of fracture healing;
* it is a dual-lag screw system that provides appropriate guidance to the sliding of the fractured extremities and an improved stability. It is effective to limit torsional instability of the femoral head, both during the intervention, by the action of tightening of the screw itself, and during the healing period due to improved bearing capacity towards multidirectional loads;
* the associated surgical instruments are simple; the low number of pieces and their ease of use made the success even of the previous version.

The aim of the present observational study is to collect data that confirm for EBA2, the technological evolution of Endovis BA, the performance and tolerability proved in the previous trial. In addition, given the increasing importance that good quality of life represents in elderly, objective of this observational study is to verify the general satisfaction of the patient with lateral proximal femoral fractures treated with EBA2.

In order to evaluate subject's walking ability after the surgical insertion of EBA2, only subjects who could walk independently before of the fracture will be included in this observational study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders, aged ≥ 60;
* Subjects with diagnosed lateral proximal femoral fractures who have undergone surgery with EBA2 nail;
* Subjects with type 31A1, 31A2 or 31A3 fractures;
* Subjects able to walk independently (with or without walking aids) before the fracture;
* Subjects who sustained a low energy injury within 72 h prior the surgery;
* Subjects who received a perioperative antibiotic therapy;
* Subjects who received antithrombotic prophylaxis for 5 weeks;
* Subjects who underwent rehabilitation procedure for 30 days at least;
* Subjects who have been mobilized in the 2nd operation day;
* Subjects able to attend the scheduled visits and to follow the instructions given by the physician;
* Subjects who have given their written informed consent.

Exclusion Criteria:

* Subjects with rheumatoid arthritis;
* Subjects with fractures due to metastasis;
* Subjects with fractures operated 72 h after the traumatic event;
* Subjects with previous ipsilateral hip or femur surgery;
* Subjects with ASA Physical Status Classification Class 5;
* Subjects with Karnofsky performance status scale before fracture ˂ 80;
* Subjects who have shown hypersensitivity to any of the components of EBA2;
* Concomitant use of any other surgical device for the femoral fracture.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone surgery with EBA2 medical device for lateral proximal femoral fracture in the period 01.08.2011 - 31.01.2012 followed by each study sites
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
EBA2 performance at day 90 | Day 90
  As a first primary endpoint, EBA2 performance will be assessed at 90 days. The performance will be assessed on the basis of failures, complications and malfunctioning related to the device.
  Since a centralized review will be performed, the extent of agreement between raters will be assessed using both Kappa statistic and AC1-statistic. Any discrepancy on the X-ray evaluation will be discussed between the raters and possibly with the Sponsor.
EBA2 performance at day 180 | Day 180
  EBA2 performance will also be assessed at 180 days. The performance will be assessed on the basis of failures, complications and malfunctioning related to the device.
EBA2 performance at day 30 (optional primary endpoint) | Day 30
  EBA2 performance will be optionally assessed at 30 days. The performance will be assessed on the basis of failures, complications and malfunctioning related to the device.

SECONDARY OUTCOMES:
SF12 Questionnaire | Day 30 (optional), 90 and 180
  The SF12 Questionnaire routinely administered to patients, will be used to assess the subjective general satisfaction of patients treated with EBA2 at day 30 (optional), 90 and 180.
Clinical evaluation of pain | Day 30 (optional), 90 and 180
  Clinical evaluation of pain data will be collected at day 30 (optional), 90 and 180 and summarized in a 4-point scale (no pain, mild, moderate, unbearable).
Radiographic examination | Day 30 (optional), 90 and 180
  The reduction maintenance, the fracture consolidation and the callus formation will be assessed through radiographic examination at day 30 (optional), 90 and 180. Frequencies and percentages will be calculated at each time point.
Walking ability data | Day 30 (optional), 90 and 180
  Walking ability data will be collected at day 30 (optional), 90 and 180 and summarized in a 3-point scale (not walking, walking with support, walking without support).
Device-related adverse events | Up to day 180
  Device-related adverse events reported during the study will be described using frequency and percentage and coded according to MedDRA coding (version 13). The number and percentage of subjects with at least one device-related adverse event will be showed. The frequency of events by SOC (System Organ Class) and PT (Preferred Term) will be reported. The characteristics of the events occurring to subjects (severity, duration, outcome, etc.) will also be summarized. The events will also be described by nature of device failure or malfunctioning.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Caiaffa, MD, Principal Investigator — S.C. Ortopedia e Traumatologia - P.O. Centrale "SS. Annunziata" ASL Taranto - Italy
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria Consorziale Policlinico, Bari
  - Unità operativa complessa di Ortopedia e Traumatologia - AUSL 12 di Viareggio, Lido di Camaiore
  - S.C. Ortopedia e Traumatologia - P.O. Centrale SS. Annunziata, Taranto

REFERENCES:
- [Background] Papasimos S, Koutsojannis CM, Panagopoulos A, Megas P, Lambiris E. A randomised comparison of AMBI, TGN and PFN for treatment of unstable trochanteric fractures. Arch Orthop Trauma Surg. 2005 Sep;125(7):462-8. doi: 10.1007/s00402-005-0021-5. PMID 16059696
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Zain Elabdien BS, Olerud S, Karlstrom G. The influence of age on the morphology of trochanteric fracture. Arch Orthop Trauma Surg (1978). 1984;103(3):156-61. doi: 10.1007/BF00435546. PMID 6497603
- [Background] Cummings SR, Nevitt MC. A hypothesis: the causes of hip fractures. J Gerontol. 1989 Jul;44(4):M107-11. doi: 10.1093/geronj/44.4.m107. PMID 2738306
- [Background] Caiaffa V, De Vita D, Laforgia R, Sessa G, Varsalona R, Girolami M, Dallari D, Mignani G, Turi G, Micaglio A, et al. Treatment of peritrochanteric fractures with the Endovis BA cephalomedullary nail: multicenter study of 1091 patients Journal of Orthopaedics and Traumatology 8(3): 111-116, 2007
- [Background] Haidukewych GJ, Israel TA, Berry DJ. Reverse obliquity fractures of the intertrochanteric region of the femur. J Bone Joint Surg Am. 2001 May;83(5):643-50. doi: 10.2106/00004623-200105000-00001. PMID 11379732
- [Background] Olsson O, Ceder L, Hauggaard A. Femoral shortening in intertrochanteric fractures. A comparison between the Medoff sliding plate and the compression hip screw. J Bone Joint Surg Br. 2001 May;83(4):572-8. doi: 10.1302/0301-620x.83b4.11302. PMID 11380135